CLINICAL TRIAL: NCT03957694
Title: A Phase 2/3 Study of AMG531 in Patients With Aplastic Anemia PreviouslyUntreated With Immunosuppressive Therapy
Brief Title: Study of AMG531(Romiplostim) in Patients With Aplastic Anemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 531-003
Record Dates: First submitted 2019-05-09; First posted 2019-05-21 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Aplastic Anemia
Keywords: aplastic anemia; romiplostim
MeSH Terms: conditions — Anemia, Aplastic | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: multi-national, open-label, phase 2/3 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMG531 (Experimental)
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Romiplostim SC. Initial dose is 10 ug/kg/. Maximum dose is 20 ug/kg. Original duration is 6 months from first administration but if investigator decide that the patient is needed more treatment, they move to extention period and take treatment up to 1 year.

SUMMARY:
To evaluate the hematological responses based on the response assessment criteria when AMG531 is subcutaneous (SC)-administered with anti-human thymocyte immunoglobulin (ATG) + ciclosporin A (CsA) therapy for 6 months in patients with aplastic anemia (AA) who were previously untreated with immunosuppressive therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signed informed consent to participate in the study;
2. A diagnosis of AA confirmed by blood and bone-marrow examinations, etc.;
3. Considered to require new treatment with ATG and CsA provided that NSAA must be platelet or erythrocyte transfusion-dependent.
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 to 1at screening

Exclusion Criteria:

1. Previously treated with ATG, CsA, or Alemtuzumab;
2. Diagnosed as having congenital AA (Fanconi anemia, congenital dyskeratosis, etc.);
3. Diagnosed as having AML or chronic myelomonocytic leukemia;
4. Concurrent thrombocytopenia of other etiologies (e.g., MDS, ITP, cirrhosis);
5. Concurrent active infection not adequately responding to appropriate therapy;
6. Concurrent clinically significant illness(es) items which are deemed by the Investigator to be likely to affect the study conduct and assessments.
7. Having active malignancies, or having a history of treatment of malignancies within 5 years prior to informed consent.
8. Concurrent PNH
9. Having Grade 2 or higher bone marrow reticulin based on Bone Marrow Pathology (2nd edition) ;
10. History of chromosome aberrations discovered in bone marrow cells.
11. Having blast cells > 2% in bone marrow;
12. Positive for anti-human immunodeficiency virus (HIV) antibody;
13. Receiving prophylactic or therapeutic treatment for hepatitis type B
14. Positive for hepatitis C virus (HCV) antibody, and HCV infection being confirmed
15. Planned hematopoietic stem cell transplantation during the study;
16. Systemic treatment with any of the following medication for the treatment of AA within 4 weeks before Day 1, however, excluding their use as premedication:

    * Anabolic steroids
    * Corticosteroids;
17. Pregnant or breastfeeding women, or women willing to become pregnant;
18. Other conditions unsuitable for participation in the study in the opinion of the Investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Achievement of complete response (CR) or partial response (PR) | 27 weeks post-dose

SECONDARY OUTCOMES:
Achievement of CR or PR | Week 14
Achievement of CR | Weeks 14 and 27
The time to CR or PR | Each time point evaluated weekly until Week 27
Reduction or independence of platelet and/or erythrocyte transfusion | Week 27
Change from baseline in platelet count (/µL) | Each time point evaluated weekly until Week 27
Change from baseline in hemoglobin (Hb) concentration (g/dL) | Each time point evaluated weekly until Week 27
Change from baseline in neutrophil count (/µL) | Each time point evaluated weekly until Week 27
Change from baseline in reticulocyte count (/µL) | Each time point evaluated weekly until Week 27

CONTACTS AND LOCATIONS:
Locations (1):
- Matsuyama Red Cross Hospital, Ehime, Japan

IPD SHARING:
Plan to Share IPD: Undecided